CLINICAL TRIAL: NCT03052725
Title: An Open-Label Extension Study of Reslizumab 110-mg Fixed, Subcutaneous Dosing in Patients 12 Years of Age and Older With Severe Eosinophilic Asthma
Brief Title: A Study of Reslizumab in Patients 12 Years of Age and Older With Severe Eosinophilic Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Parent Studies didn't meet their primary endpoint so study was terminated.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C38072-AS-30066; 2016-004661-23 (EudraCT Number)
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Results first posted 2019-03-21 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Eosinophils, Asthma
MeSH Terms: conditions — Asthma | interventions — reslizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- reslizumab 110 mg (Experimental): Reslizumab was administered as 110 mg subcutaneous (sc) injection in the thigh, abdomen, or upper arm(s) once every 4 weeks for a total of 9 doses.
  Interventions: Drug: reslizumab

INTERVENTIONS:
Drug: reslizumab — Reslizumab was provided in a pre-filled syringe.
  Other Names: CEP38072

SUMMARY:
This is a multicenter, open-label (OL) extension study to obtain additional long-term safety data for subcutaneous (sc) administration of reslizumab treatment administered at a fixed dose of 110 mg in patients 12 years of age and older with severe eosinophilic asthma who completed the treatment period of a placebo-controlled Phase 3 trial of sc reslizumab. The study consists of a screening/baseline visit followed by a 36-week OL treatment period and a 15-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

• Patient with eosinophilic asthma who completed the treatment period of a double-blind, placebo controlled sc reslizumab study (Study C38072-AS-30025 or C38072-AS-30027)

~~ Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Patient has received any reslizumab administration in any previous clinical trial other than Studies C38072-AS-30025 and C38072-AS-30027.
* The patient has any clinically significant, uncontrolled medical condition
* The patient has another confounding underlying lung disorder
* The patient has a known/diagnosed hypereosinophilic syndrome.
* The patient has a diagnosis of malignancy within 5 years of the screening visit, except for treated and cured non-melanoma skin cancers.
* The patient is a pregnant or lactating woman
* The patient is a current smoker (ie, has smoked within the last 6 months before screening) or has a smoking history ≥10 pack-years.
* The patient is currently using any systemic immunosuppressive or immunomodulatory agents other than OCS
* The patient has a history of allergic reaction or hypersensitivity to any component of the study drug.
* The patient has a history of an immunodeficiency disorder including human immunodeficiency virus (HIV).

  * Additional criteria apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (134):
- United States (37):
  - Teva Investigational Site 14647, Birmingham, Alabama
  - Teva Investigational Site 14631, Bakersfield, California
  - Teva Investigational Site 14648, Huntington Beach, California
  - Teva Investigational Site 14637, Napa, California
  - Teva Investigational Site 14654, Stockton, California
  - Teva Investigational Site 14636, Walnut Creek, California
  - Teva Investigational Site 14626, Aventura, Florida
  - Teva Investigational Site 14634, Homestead, Florida
  - Teva Investigational Site 14650, Miami, Florida
  - Teva Investigational Site 14629, Miami, Florida
  - Teva Investigational Site 14619, Miami, Florida
  - Teva Investigational Site 14624, Orlando, Florida
  - Teva Investigational Site 14638, Tallahassee, Florida
  - Teva Investigational Site 14642, Buford, Georgia
  - Teva Investigational Site 14651, Chicago, Illinois
  - Teva Investigational Site 14645, Michigan City, Indiana
  - Teva Investigational Site 14620, Owensboro, Kentucky
  - Teva Investigational Site 14623, Lafayette, Louisiana
  - Teva Investigational Site 14627, North Dartmouth, Massachusetts
  - Teva Investigational Site 14644, Boys Town, Nebraska
  - Teva Investigational Site 14652, Ocean City, New Jersey
  - Teva Investigational Site 14632, Lake Success, New York
  - Teva Investigational Site 14646, New York, New York
  - Teva Investigational Site 14633, Cincinnati, Ohio
  - Teva Investigational Site 14653, Cleveland, Ohio
  - Teva Investigational Site 14621, Edmond, Oklahoma
  - Teva Investigational Site 14625, Edmond, Oklahoma
  - Teva Investigational Site 14643, Jenkintown, Pennsylvania
  - Teva Investigational Site 14622, Pittsburgh, Pennsylvania
  - Teva Investigational Site 14630, East Providence, Rhode Island
  - Teva Investigational Site 14649, Providence, Rhode Island
  - Teva Investigational Site 14655, Knoxville, Tennessee
  - Teva Investigational Site 14639, Corsicana, Texas
  - Teva Investigational Site 14640, Dallas, Texas
  - Teva Investigational Site 14641, Provo, Utah
  - Teva Investigational Site 14628, Abingdon, Virginia
  - Teva Investigational Site 14635, Falls Church, Virginia
- Belgium (3):
  - Teva Investigational Site 37082, Brussels
  - Teva Investigational Site 37081, Erpent
  - Teva Investigational Site 37083, Ghent
- Canada (2):
  - Teva Investigational Site 11133, Vancouver, British Columbia
  - Teva Investigational Site 11134, Etobicoke, Ontario
- Czechia (4):
  - Teva Investigational Site 54151, Břeclav
  - Teva Investigational Site 54150, Jablonec nad Nisou
  - Teva Investigational Site 54148, Jindřichův Hradec
  - Teva Investigational Site 54149, Tábor
- France (3):
  - Teva Investigational Site 35229, Le Kremlin-Bicêtre
  - Teva Investigational Site 35227, Strasbourg
  - Teva Investigational Site 35228, Toulouse
- Germany (13):
  - Teva Investigational Site 32670, Berlin
  - Teva Investigational Site 32680, Berlin
  - Teva Investigational Site 32673, Berlin
  - Teva Investigational Site 32679, Frankfurt
  - Teva Investigational Site 32675, Frankfurt am Main
  - Teva Investigational Site 32678, Hamburg
  - Teva Investigational Site 32681, Hanover
  - Teva Investigational Site 32677, Koblenz
  - Teva Investigational Site 32672, Leipzig
  - Teva Investigational Site 32671, Leipzig
  - Teva Investigational Site 32674, Lübeck
  - Teva Investigational Site 32682, Rostock
  - Teva Investigational Site 32676, Tempelhof
- Hungary (14):
  - Teva Investigational Site 51291, Balassagyarmat
  - Teva Investigational Site 51290, Budapest
  - Teva Investigational Site 51293, Csorna
  - Teva Investigational Site 51292, Debrecen
  - Teva Investigational Site 51283, Debrecen
  - Teva Investigational Site 51286, Gödöllő
  - Teva Investigational Site 51284, Győr
  - Teva Investigational Site 51285, Hajdúnánás
  - Teva Investigational Site 51282, Kapuvár
  - Teva Investigational Site 51288, Szeged
  - Teva Investigational Site 51289, Szigetvár
  - Teva Investigational Site 51280, Szombathely
  - Teva Investigational Site 51281, Tatabánya
  - Teva Investigational Site 51287, Veszprém
- Israel (8):
  - Teva Investigational Site 80136, Ashkelon
  - Teva Investigational Site 80129, Haifa
  - Teva Investigational Site 80131, Jerusalem
  - Teva Investigational Site 80135, Jerusalem
  - Teva Investigational Site 80134, Kfar Saba
  - Teva Investigational Site 80132, Petah Tikva
  - Teva Investigational Site 80133, Ramat Gan
  - Teva Investigational Site 80130, Rehovot
- Poland (10):
  - Teva Investigational Site 53405, Bialystok
  - Teva Investigational Site 53402, Gdansk
  - Teva Investigational Site 53399, Krakow
  - Teva Investigational Site 53408, Lodz
  - Teva Investigational Site 53400, Lodz
  - Teva Investigational Site 53403, Lubin
  - Teva Investigational Site 53407, Ostrów Wielkopolski
  - Teva Investigational Site 53401, Poznan
  - Teva Investigational Site 53404, Tarnów
  - Teva Investigational Site 53406, Wroclaw
- Romania (5):
  - Teva Investigational Site 52115, Brasov
  - Teva Investigational Site 52116, Brasov
  - Teva Investigational Site 52113, Cluj-Napoca
  - Teva Investigational Site 52114, Târgu Mureş
  - Teva Investigational Site 52117, Timișoara
- Russia (9):
  - Teva Investigational Site 50460, Barnaul
  - Teva Investigational Site 50453, Kemerovo
  - Teva Investigational Site 50461, Kemerovo
  - Teva Investigational Site 50456, Moscow
  - Teva Investigational Site 50459, Moscow
  - Teva Investigational Site 50455, Novosibirsk
  - Teva Investigational Site 50454, Saint Petersburg
  - Teva Investigational Site 50457, Saint Petersburg
  - Teva Investigational Site 50458, Tomsk
- Spain (3):
  - Teva Investigational Site 31219, Barcelona
  - Teva Investigational Site 31218, Valencia
  - Teva Investigational Site 31217, Valencia
- Ukraine (23):
  - Teva Investigational Site 58283, Chernivtsi
  - Teva Investigational Site 58304, Dnipropetrovsk
  - Teva Investigational Site 58287, Dnipropetrovsk
  - Teva Investigational Site 58295, Ivano-Frankivsk
  - Teva Investigational Site 58293, Kharkiv
  - Teva Investigational Site 58289, Kharkiv
  - Teva Investigational Site 58284, Kharkiv
  - Teva Investigational Site 58288, Kharkiv
  - Teva Investigational Site 58302, Kremenchuk
  - Teva Investigational Site 58292, Kryvyi Rih
  - Teva Investigational Site 58303, Kyiv
  - Teva Investigational Site 58282, Kyiv
  - Teva Investigational Site 58285, Kyiv
  - Teva Investigational Site 58286, Kyiv
  - Teva Investigational Site 58290, Kyiv
  - Teva Investigational Site 58291, Kyiv
  - Teva Investigational Site 58296, Kyiv
  - Teva Investigational Site 58299, Kyiv
  - Teva Investigational Site 58297, Sumy
  - Teva Investigational Site 58294, Vinnytsia
  - Teva Investigational Site 58301, Vinnytsia
  - Teva Investigational Site 58298, Zaporizhzhya
  - Teva Investigational Site 58300, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 392 patients with severe eosinophilic asthma rolled over from Study 30025 or 30027, and 391 of these patients (at 125 centers) were enrolled into this extension study and treated with reslizumab. One patient withdrew consent after completing Study 30025 and before enrolling in Study 30066.
Pre-assignment Details: Of the 391 patients enrolled, 112 (29%) enrolled seamlessly and 279 (71%) enrolled non-seamlessly, meaning there was a time gap between completion of the parent study and start of this extension study.
Groups:
- Reslizumab 110 mg; Previous Treatment Placebo: Participants who were administered placebo in the parent study, were administered reslizumab 110 mg by subcutaneous injection every 4 weeks for a total of 9 doses.
- Reslizumab 110 mg: Previous Treatment Reslizumab: Participants who were administered reslizumab in the parent study, were administered reslizumab 110 mg by subcutaneous injection every 4 weeks for a total of 9 doses.
Period: Overall Study
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg: Previous Treatment Reslizumab
Started | 194 | 197
Safety Analysis Set (Enrolled and treated) | 194 | 196
Completed (Completed treatment; due to study termination, the end of study visit was not conducted.) | 46 | 47
Not Completed | 148 | 150
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Pregnancy | 0 | 1
Not completed — Site closure | 0 | 1
Not completed — Study terminated by sponsor | 143 | 144

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg: Previous Treatment Reslizumab | Total
Number analyzed (Participants) | 194 | 197 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (14.85) | 52.5 (15.62) | 51.5 (15.26)
Age, Customized [Count of Participants; unit: Participants]
  12 to <18 years | 9 | 8 | 17
  18 to <65 years | 156 | 141 | 297
  >=65 years | 29 | 48 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 122 | 234
  Male | 82 | 75 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 8 | 26
  Not Hispanic or Latino | 174 | 187 | 361
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 182 | 185 | 367
    Black | 7 | 10 | 17
    Asian | 3 | 2 | 5
    Other | 2 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] — Population: Some participants were missing a baseline weight measurement.
  kg
    number analyzed (Participants) | 186 | 184 | 370
    (all) | 79.78 (17.647) | 81.22 (18.712) | 80.49 (18.174)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Some participants were missing a baseline BMI measure.
  kg/m^2
    number analyzed (Participants) | 184 | 182 | 366
    (all) | 28.377 (5.8288) | 28.880 (5.9672) | 28.627 (5.8954)
Systemic Corticosteroid (OCS) Use at Baseline [Mean (Standard Deviation); unit: mg prednisolone or equivalent] — Daily OCS dose is defined as total OCS dose in a day (accounting for reported dose and dose frequency) and converting the total daily dose to a prednisone-equivalent dose. Population: Safety Analysis set of participants on daily OCS at baseline
  mg prednisolone or equivalent
    number analyzed (Participants) | 46 | 45 | 91
    (all) | 12.01 (10.870) | 12.26 (10.760) | 12.14 (10.756)
Region Group [Count of Participants; unit: Participants] — Population: Enrolled analysis set
  Participants
    U.S./Canada | 47 | 41 | 88
    Europe | 131 | 136 | 267
    Other | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence, regardless of whether it has a causal relationship with study treatment. In this study, asthma exacerbations should not be recorded as adverse events unless assessed by the investigator as more severe than the patient's usual disease course. The period for reporting treatment-emergent adverse events was defined as the period after the first dose of study drug was administered until the end of treatment visit. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to up to Day 269; for participants who discontinued early for reasons other than study termination, the timeframe was first dose of study drug to 4 weeks after the last dose of study drug.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Reslizumab 110 mg; Previous Treatment Reslizumab: Participants who were administered reslizumab in the parent study, were administered reslizumab 110 mg by subcutaneous injection every 4 weeks for a total of 9 doses.
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
Participants
  >=1 TEAE | 102 | 114
  >=1 treatment-related TEAE | 7 | 6
  >=1 serious TEAE | 5 | 11
  >=1 treatment-related, serious TEAE | 0 | 0
  >=1 TEAE leading to discontinuation | 2 | 0
  >=1 TEAE leading to death | 0 | 0

2. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Hematology Values
Description: Participants are included in the counts if the worst study value reaches the following clinically significant levels:
  Eosinophils (high): >=1.5*10^9/L and increase >0 Hematocrit (low): >=18 years old: <0.32 L/L for females; <0.37 L/L for males plus a decrease >0 for both or 12 to <18 years old: <0.30 L/L and a decrease >0 for both females and males Hemoglobin (low): >=18 years old: <=95 g/L and decrease >0; 12 to <18 years old: <=100 g/L and decrease >0 Leukocytes (high): >=20*10^9/L and increase >0 Leukocytes (low): <=3*10^9/L and decrease >0 Neutrophils (low): <=1*10^9/L and decrease >0 Platelets (low): <=75*10^9/L and decrease >0
Time Frame: Week 0 (baseline), Weeks 8, 24, 36 plus any unscheduled visits
Population: Safety analysis set of participants with a baseline and post-baseline result for each variable
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 192 | 192
Participants
  Participants with >=1 abnormality | 8 | 5
  Eosinophils (high): number analyzed (Participants) | 191 | 192
  Eosinophils (high) | 1 | 0
  Hematocrit (low) | 4 | 2
  Hemoglobin (low) | 2 | 0
  Leukocytes (high) | 0 | 1
  Leukocytes (low) | 2 | 0
  Neutrophils (low): number analyzed (Participants) | 191 | 192
  Neutrophils (low) | 1 | 1
  Platelets: number analyzed (Participants) | 190 | 189
  Platelets | 0 | 1

3. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Serum Chemistry Values
Description: Participants are included in the counts if the worst study value reaches the following clinically significant levels:
  Alanine Aminotransferase (high): >=3* upper limit of normal (ULN) and increase >0 Aspartate Aminotransferase (high): >=3* upper limit of normal (ULN) and increase >0 Bilirubin (high): >=34.2 micromol/L and increase >0 Blood Urea Nitrogen (high): >=10.71 mmol/L and increase >0 Creatine Phosphokinase (high): >10* ULN and increase >0 Creatine Phosphokinase (medium high): >=3.1*ULN and <=10*ULN and increase >0 Creatinine (high): >=177 micromol/L and increase >0
Time Frame: Week 0 (baseline), Weeks 4, 8, 24, 36 plus any unscheduled visits
Population: Safety analysis set of participants with a baseline and post-baseline result for each variable
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 193 | 192
Participants
  Participants with >=1 abnormality | 12 | 10
  Alanine Aminotransferase (high) | 1 | 2
  Aspartate Aminotransferase (high) | 1 | 1
  Bilirubin (high) | 2 | 1
  Blood Urea Nitrogen (high) | 2 | 4
  Creatine Phosphokinase (high) | 2 | 1
  Creatine Phosphokinase (medium high) | 6 | 4
  Creatinine (high) | 0 | 1

4. Secondary Outcome: Participants' Tolerability and Injection Site Reactions by Domain and Worst Overall Severity
Description: The worst finding for participants in each tolerability and injection site domain from all treatment weeks is summarized. Local tolerability at the injection site was assessed approximately 1 hour after study drug administration.
  Severity was rated on a 4-level scale of none, mild, moderate and severe.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, and 36
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
Participants
  Pain - None | 191 | 194
  Pain - Mild | 3 | 2
  Pain - Moderate | 0 | 0
  Pain - Severe | 0 | 0
  Tenderness - None | 193 | 192
  Tenderness - Mild | 1 | 4
  Tenderness - Moderate | 0 | 0
  Tenderness - Severe | 0 | 0
  Erythema - None | 191 | 188
  Erythema - Mild | 2 | 7
  Erythema - Moderate | 1 | 1
  Erythema - Severe | 0 | 0
  Warmth - None | 192 | 192
  Warmth - Mild | 1 | 4
  Warmth - Moderate | 1 | 0
  Warmth - Severe | 0 | 0
  Swelling - None | 191 | 190
  Swelling - Mild | 2 | 5
  Swelling - Moderate | 1 | 1
  Swelling - Severe | 0 | 0

5. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Sign Values
Description: Participants are included in the counts if the worst study value reaches the following clinically significant levels:
  Diastolic blood pressure (high): >100 mmHg and increase >=12 for participants >=18 years; >85 mmHg and increase >=12 for participants 12 - < 18 years Pulse rate (high): >100 beats/minute and increase >=12 Respiratory rate (high): >24 breaths/minute and increase >=10 for participants >=18 years >20 breaths/minute and increase >=10 for participants 12 - < 18 years Systolic blood pressure (high): >160 mmHg and increase >=30 for participants >=18 years; >130 mmHg and increase >=30 for participants 12 - < 18 years Temperature (high): >38.1 celsius and increase >=1.1 Temperature (low): <35.8 celsius
Time Frame: Week 0 (baseline), Weeks 4, 8, 12, 16,20, 24, 28, 32, 36 plus any unscheduled visits
Population: Safety analysis set of participants with a baseline and post-baseline result for each variable
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 193 | 196
Participants
  Participants with >=1 abnormality | 20 | 16
  Diastolic Blood Pressure - High | 0 | 1
  Pulse Rate - High | 1 | 2
  Respiratory Rate - High | 2 | 0
  Systolic Blood Pressure - High | 2 | 0
  Temperature - High | 1 | 0
  Temperature - Low | 14 | 13

6. Secondary Outcome: Annualized Rate of Clinical Asthma Exacerbations (CAEs)
Description: Data is included between the first dose of study drug to the end of treatment visit for completed participants, and the first dose of study drug to 4 weeks after the last dose of study drug for patients who discontinued treatment early.
  Annual rate is defined as the number of events/(duration of treatment [days]/365.25).
  Participants with zero events are included.
Time Frame: as for outcome 1
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: CAEs / year
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
CAEs / year | 0.42 (1.104) | 0.70 (1.538)

7. Secondary Outcome: Annualized Rate of Clinical Asthma Exacerbations (CAEs) Requiring Asthma-Specific Hospital Admissions or Emergency Room Visits
Description: as for outcome 6
Time Frame: as for outcome 1
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: CAEs / year
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
CAEs / year | 0.06 (0.362) | 0.11 (0.514)

8. Secondary Outcome: Mean Number of Days of Hospital Stay During the Treatment Period
Description: Participants with no hospitalizations are included.
Time Frame: as for outcome 1
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
days | 0.25 (1.658) | 1.02 (7.848)

9. Secondary Outcome: Mean Number of School/Work Days Missed Due to Asthma During the Treatment Period
Description: Participants with no school or work days missed due to asthma are included in the counts.
Time Frame: as for outcome 1
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
days | 0.11 (1.202) | 0.00 (0.000)

10. Secondary Outcome: Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1): Baseline Values and Change From Baseline Values at Weeks 8, 24 and 36
Description: The FEV1 is the volume of air that can be forcibly exhaled from the lungs in the first second, measured in liters.
  Pre-bronchodilator spirometry assessments at designated clinic visits (weeks 0, 8, and 24, and 36) should only be performed after withholding short-acting bronchodilators (ie, inhaled short-acting beta-adrenergic agonists and/or short-acting anticholinergics) for at least 6 hours and long-acting bronchodilators ie, inhaled long-acting beta-adrenergic agonists and long acting anticholinergic agents) for at least 12 or 24 hours, according to their labeled dose schedule.
Time Frame: Week 0 (baseline), Weeks 8, 24, 36
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
liters
  Baseline - observed value: number analyzed (Participants) | 179 | 177
  Baseline - observed value | 2.162 (0.980) | 2.117 (0.927)
  Change at Week 8: number analyzed (Participants) | 175 | 168
  Change at Week 8 | 0.099 (0.704) | 0.031 (0.529)
  Change at Week 24: number analyzed (Participants) | 99 | 91
  Change at Week 24 | 0.169 (0.851) | -0.020 (0.472)
  Change at Week 36: number analyzed (Participants) | 32 | 31
  Change at Week 36 | 0.245 (0.677) | 0.010 (0.550)

11. Secondary Outcome: Morning Ambulatory Forced Expiratory Volume in One Second (FEV1): Baseline Values and Change From Baseline Values at Weeks 1, 4, 8, 24 and 36
Description: A weekly average of daily morning ambulatory FEV1 (measured by the handheld spirometry device) was derived using 7-day window intervals. The average was calculated as the sum of all values divided by the number of non-missing assessments. There will be no imputation of missing data. At least 4 of the 7 measurements need to be recorded for a week to be included in the analysis; otherwise the week was treated as missing.
Time Frame: Week 0 (baseline), Weeks 1, 4, 8, 24, 36
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
liters
  Baseline - observed value: number analyzed (Participants) | 192 | 193
  Baseline - observed value | 2.057 (0.814) | 2.027 (0.847)
  Change at Week 1: number analyzed (Participants) | 190 | 186
  Change at Week 1 | 0.002 (0.345) | -0.044 (0.291)
  Change at Week 4: number analyzed (Participants) | 184 | 190
  Change at Week 4 | 0.051 (0.490) | -0.049 (0.319)
  Change at Week 8: number analyzed (Participants) | 185 | 187
  Change at Week 8 | 0.028 (0.463) | -0.039 (0.345)
  Change at Week 24: number analyzed (Participants) | 150 | 146
  Change at Week 24 | 0.051 (0.492) | -0.062 (0.403)
  Change at Week 36: number analyzed (Participants) | 33 | 34
  Change at Week 36 | 0.061 (0.273) | -0.053 (0.465)

12. Secondary Outcome: Percent Change From Baseline in Daily Oral Corticosteroid (OCS) Dose During Weeks 16-20 and Weeks 32-36
Description: Daily OCS dose is defined as total OCS dose in a day (accounting for reported dose and dose frequency) and converting the total daily dose to a prednisone-equivalent dose.
  Baseline dose is the prescribed OCS dose on the day of first dose of study drug in this study. Dose at Weeks 16-20 and 32-36 is the mean of all daily OCS doses during the week range.
  Percent change = 100 * (absolute change / baseline dose)
Time Frame: Week 0 (baseline), Weeks 16-20, Weeks 32-36
Population: Safety Analysis set of participants on daily OCS at baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 46 | 45
percent change
  % change at Week 16-20 | -2.19 (51.347) | -6.96 (40.904)
  % change at Week 32-36: number analyzed (Participants) | 11 | 11
  % change at Week 32-36 | -8.44 (24.236) | -8.75 (29.666)

13. Secondary Outcome: Total Inhalations of Reliever Bronchodilator Medication: Baseline Values and Change From Baseline Values at Weeks 1, 4, 8, 24 and 36
Description: Total inhalations of reliever bronchodilator medication (eg, short-acting beta-agonist [SABA]) measured using weekly averages.
  The average was calculated as the sum of all values divided by the number of non-missing assessments. There was no imputation of missing data. At least 4 of the 7 measurements need to be recorded for a week to be included in the analysis; otherwise the week was treated as missing.
Time Frame: Baseline (Week 0), Weeks 1, 4, 8, 24, 36
Population: Safety Analysis set
Measure: Mean (Standard Deviation); unit: inhalations
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
inhalations
  Baseline - observed values: number analyzed (Participants) | 171 | 170
  Baseline - observed values | 2.4 (3.39) | 2.6 (3.10)
  Change at Week 1: number analyzed (Participants) | 158 | 160
  Change at Week 1 | -0.4 (1.30) | -0.4 (1.17)
  Change at Week 4: number analyzed (Participants) | 153 | 162
  Change at Week 4 | -0.6 (1.86) | -0.5 (1.50)
  Change at Week 8: number analyzed (Participants) | 155 | 163
  Change at Week 8 | -0.7 (1.79) | -0.6 (1.61)
  Change at Week 24: number analyzed (Participants) | 121 | 118
  Change at Week 24 | -0.8 (1.92) | -0.8 (1.78)
  Change at Week 36: number analyzed (Participants) | 23 | 25
  Change at Week 36 | -0.5 (1.69) | -0.6 (1.80)

14. Secondary Outcome: Asthma Control Questionnaire-6 (ACQ-6) Total Score: Baseline Values and Change From Baseline Values at Weeks 8, 24 and 36
Description: The ACQ-6 is a validated asthma assessment tool that has been widely used. There are 6 self-assessment questions. Each item on the ACQ-6 has a possible score ranging from 0 to 6 and the total score is the mean of all responses. The seven-point response scale: 0 = 'totally controlled' and 6 = 'severely uncontrolled.' Negative change from baseline values indicate improved asthma control.
Time Frame: Baseline (Week 0), Weeks 8, 24, 36
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
units on a scale
  Baseline - observed values: number analyzed (Participants) | 193 | 195
  Baseline - observed values | 1.72 (1.098) | 1.69 (1.171)
  Change at Week 8: number analyzed (Participants) | 191 | 192
  Change at Week 8 | -0.31 (0.777) | -0.20 (0.718)
  Change at Week 24: number analyzed (Participants) | 150 | 145
  Change at Week 24 | -0.30 (0.936) | -0.23 (0.771)
  Change at Week 36: number analyzed (Participants) | 78 | 77
  Change at Week 36 | -0.34 (0.855) | -0.28 (0.867)

15. Secondary Outcome: Asthma Quality of Life Questionnaire Administered to Participants Ages 12-70 Years (AQLQ +12) Overall Score: Baseline Values and Change From Baseline Values at Weeks 8, 24 and 36
Description: The AQLQ +12 is a modified version of the standardized AQLQ, which was developed to measure functional impairments experienced by adults ≥17 years of age. The AQLQ +12 is valid for patients 12 to 70 years of age and includes 32 questions in 4 domains (symptoms, activity limitation, emotional function, and environmental stimuli). Participants were asked to recall their experiences during the previous 2 weeks and score each of the questions on a 7-point scale, where 7=not at all limited and 1=totally limited. The overall score of the AQLQ +12 was derived as the average of the 32 questions, thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment").
  Positive change from baseline values indicate improved quality of life.
Time Frame: Baseline (Week 0), Weeks 8, 24, 36
Population: Safety Analysis set of participants age 12-70 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 187 | 179
units on a scale
  Baseline - observed value: number analyzed (Participants) | 186 | 176
  Baseline - observed value | 5.04 (1.249) | 5.14 (1.270)
  Change at Week 8: number analyzed (Participants) | 185 | 173
  Change at Week 8 | 0.30 (0.716) | 0.14 (0.700)
  Change at Week 24: number analyzed (Participants) | 143 | 131
  Change at Week 24 | 0.28 (0.727) | 0.20 (0.830)
  Change at Week 36: number analyzed (Participants) | 72 | 68
  Change at Week 36 | 0.32 (0.835) | 0.19 (0.948)

16. Secondary Outcome: Participants With Treatment-Emergent Anti-Drug Antibody (ADA) Responses
Description: Treatment-emergent responses were defined as a positive sample post-baseline (negative baseline) OR a titer increase of >=4-fold relative to a positive baseline sample.
  Two types of antibody assay were performed, an immunogenicity status assay (ADA) and neutralizing assay (NAb).
  The ADA assay produces a positive or negative result. For samples with a positive result, a neutralizing assay was performed, which also produces a positive or negative result.
Time Frame: Baseline - date of randomization in the previous study (C38072-AS-30025 or C38072-AS-30027), Weeks 8, 24, 36 or early withdrawal
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 194 | 196
Participants | 11 | 9

17. Secondary Outcome: Participants With Treatment-Emergent Anti-Drug Antibody (ADA) At the End-0f-Study Visit (Week 51)
Description: The endpoint was defined to evaluate immunogenicity after study drug washout since the end of study visit on Week 51 was to be 19 weeks after the final dose of study drug. Due to the early termination of the study no participants had an end of study visit.
Time Frame: Week 51
Population: Safety Analysis set
Arm/Group | Reslizumab 110 mg; Previous Treatment Placebo | Reslizumab 110 mg; Previous Treatment Reslizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to up to Day 269; for participants who discontinued early for reasons other than study termination, the timeframe was first dose of study drug to 4 weeks after the last dose of study drug.
Groups:
- Reslizumab 110 mg: Participants were administered reslizumab 110 mg by subcutaneous injection every 4 weeks for a total of 9 doses.
Arm/Group | Reslizumab 110 mg
All-Cause Mortality (participants affected / at risk) | 0/390
Serious Adverse Events (participants affected / at risk) | 16/390
Other Adverse Events (participants affected / at risk) | 70/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 110 mg (N=390)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 110 mg (N=390)
Upper respiratory tract infection (Infections and infestations) | 23 (24)
Viral upper respiratory tract infection (Infections and infestations) | 49 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03052725/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT03052725/SAP_001.pdf